CLINICAL TRIAL: NCT01225172
Title: A Phase 2 Study of BMS-754807 Combined With Letrozole or BMS-754807 Alone in Hormone Receptor-Positive Breast Cancer Subjects With Acquired Resistance to Non-Steroidal Aromatase Inhibitors
Brief Title: Study of BMS-754807 Combined With Letrozole or BMS-754807 Alone in Patients With Hormone Receptor-Positive Breast Cancer and Resistance to Non-Steroidal Aromatase Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA191-011
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BMS 754807; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-754807 (Experimental)
  Interventions: Drug: BMS-754807
- BMS-754807 + letrozole (Experimental)
  Interventions: Drug: BMS-754807; Drug: letrozole

INTERVENTIONS:
Drug: BMS-754807 — Tablet, Oral, 100 mg, Daily, Until disease progression or unacceptable toxicity
Drug: letrozole — Tablets, Oral, 2.5 mg, Daily, Until disease progression or unacceptable toxicity
  Other Names: Femara®
  Arms: BMS-754807 + letrozole

SUMMARY:
The purpose of this study is to evaluate oral doses of BMS-754807 in combination with letrozole or BMS-754807 alone are safe and efficacious in locally advanced or metastatic hormone receptor positive breast cancer subjects who have progressed with prior non-steroidal aromatase inhibitor treatment.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Postmenopausal women with hormone receptor-positive and HER-2 negative breast cancer
* Disease progression following non-steroidal aromatase inhibitor treatment

Exclusion Criteria:

* Known symptomatic brain metastasis
* Medical condition requiring chronic steroids
* History of Type 1 or 2 Diabetes
* Uncontrolled or significant cardiovascular (CV) disease
* Concomitant second malignancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-12-31 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (17):
  - Univ Of Al At Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Sharp Clinical Oncology Research, San Diego, California
  - Mayo Clinic, Jacksonville, Florida
  - University Of Chicago Medical Center, Chicago, Illinois
  - Illinois Cancercare, Pc, Peoria, Illinois
  - Indiana University Health Goshen Center For Cancer Care, Goshen, Indiana
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Oncology Care Associates, P.A., Wheaton, Maryland
  - Masonic Cancer Ctr, University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Unv. Of Nc At Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Hospital Cancer Research, Charlotte, North Carolina
  - Duke University Medical Center-Dept Of Medicine, Durham, North Carolina
  - Ut Md Anderson Can Ctr., Houston, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - University Of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 participants were enrolled, 59 of whom were treated. Reasons for not entering treatment period included: 3 participants withdrew consent; 11 participants no longer met study criteria and 4 were due to other reasons.
Groups:
- BMS 100+LET: Treatment with 100 mg BMS-754807 + 2.5 mg letrozole
- BMS 100: 100 mg BMS-754807 alone
Period: Overall Study
Arm/Group | BMS 100+LET | BMS 100
Started | 52 | 7
Completed | 46 | 6
Not Completed | 6 | 1
Not completed — Subject decision to stop | 1 | 0
Not completed — Subject request to discontinue treatment | 3 | 1
Not completed — Subject no longer meets study criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS 100+LET | BMS 100 | Total
Number analyzed (Participants) | 52 | 7 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 4 | 39
  >=65 years | 17 | 3 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (12.21) | 64.4 (8.58) | 60.5 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 7 | 59
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 50 | 6 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 46 | 6 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 24 Weeks
Description: Progression free survival (PFS) rate at 24 weeks after treatment with BMS 754807/letrozole was to be calculated as the total number of subjects neither progressed nor died after 24 weeks of treatment divided by the total number of subjects (with measurable or non-measurable disease) randomized/assigned to combination treatment arm and treated. In participants with measurable disease Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) criteria was to be used to assess disease progression.This outcome was not measured due to early termination of the study.
Time Frame: 24 weeks after initiation of study treatment
Population: PFS data was not collected for any participants because the study was terminated
Groups:
- BMS 100 + LET: Treatment with 100 mg BMS-754807 + 2.5 mg letrozole
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Objective Response Rate (ORR) in Participants With Measurable Disease
Description: ORR is defined as the number of participants with best overall response (OR) of confirmed complete response (CR) or partial response (PR) divided by the number of participants who received treatment.
  Participants were to be evaluated for tumor response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions.: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. This outcome measure was not met due to early termination of the study
Time Frame: 24 weeks after initiation of study treatment
Population: ORR data was not collected for any participants because the study was terminated
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, Non-serious AEs , Discontinuation Due to AEs and Deaths
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment.
Time Frame: Non-SAEs: Day 1 to 7 days after the participant discontinues study medication or 7 days after the End of Treatment visit (up to 42 months), For SAEs: during the screening period and within 30 days of discontinuation of dosing ,up to 42 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 52 | 7
Participants
  No. of deaths | 5 | 0
  No. of participants with Serious AEs | 11 | 1
  No. of participants with AEs (All grades) | 51 | 7
  No. of discontinuations due to AEs | 11 | 2
  No. of participants with non-serious AEs | 51 | 7

4. Secondary Outcome: Duration of Response (DOR) in Participants With Measurable Disease
Description: DOR was to be performed to further characterize the response rate at Week 24. Duration of response is defined as the time between the Week 25 date of response and the date of objectively documented disease progression as defined by modified RECIST 1.1 criteria or death, whichever occurs first. DOR could not be assessed due to early termination of the study.
Time Frame: 24 weeks after initiation of study treatment
Population: DOR data was not collected for any participants because the study was terminated early
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of On-study Laboratory Abnormalities: Grade 1-2
Description: Blood and urine samples were obtained at specified times points for laboratory evaluations. Clinical Laboratory Sage Panels included: Hematology: Hemoglobin, Hematocrit, Red blood cell, Total leukocyte count, including differential, Platelet count. Serum Chemistry : Albumin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALK-P), Bilirubin, total (TB). Reflex testing of direct (conjugated) and indirect (unconjugated) bilirubin will be ordered if total bilirubin > 5X ULN, Blood urea nitrogen (BUN or urea), Calcium, Chloride, Cholesterol, Creatinine, serum, Glucose, fasting plasma, Lactate dehydrogenase (LDH), Magnesium, Phosphorus, Potassium, Protein, total, Sodium, Triglycerides, Uric acid Urinalysis, Blood, Glucose, Ketones, Leukocyte esterase, pH, Protein. Laboratory tests were graded using the National Cancer Institute-Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0 criteria
Time Frame: Assessed from day 1 up to within 30 days of last dose (Approximately 42 months)
Population: All treated participants
Measure: Number; unit: Number of abnormalities
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 52 | 7
Number of abnormalities
  Albumin | 13 | 0
  Alkaline Phosphatase (ALP) | 12 | 2
  Alanine Aminotransferase (ALT) | 7 | 1
  Aspartate Aminotransferase (AST) | 17 | 1
  Cholesterol, Total (TC): number analyzed (Participants) | 50 | 7
  Cholesterol, Total (TC) | 28 | 4
  Creatinine | 11 | 0
  Absolute Neutrophil Count | 16 | 3
  Hemoglobin | 27 | 1
  Lymphocytes (absolute) | 32 | 4
  Magnesium , serum: number analyzed (Participants) | 51 | 7
  Magnesium , serum | 13 | 1
  Neutrophils (absolute): number analyzed (Participants) | 51 | 7
  Neutrophils (absolute) | 15 | 2
  Glucose, fasting plasma: number analyzed (Participants) | 43 | 7
  Glucose, fasting plasma | 21 | 3
  Phosphorus, inorganic: number analyzed (Participants) | 51 | 7
  Phosphorus, inorganic | 5 | 0
  Platelet count | 14 | 1
  Bilirubin, total | 3 | 1
  Triglycerides: number analyzed (Participants) | 37 | 7
  Triglycerides | 1 | 0
  Triglycerides, fasting: number analyzed (Participants) | 42 | 7
  Triglycerides, fasting | 15 | 2
  Uric acid: number analyzed (Participants) | 51 | 7
  Uric acid | 10 | 1
  Leukocytes | 17 | 3

6. Secondary Outcome: Number of On-study Laboratory Abnormalities: Grade 3-4
Description: Blood and urine samples were obtained at specified times points for laboratory evaluations. Clinical Laboratory Sage Panels included: Hematology: Hemoglobin, Hematocrit, Red blood cell, Total leukocyte count, including differential, Platelet count. Serum Chemistry : Albumin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALK-P), Bilirubin, total (TB). Reflex testing of direct (conjugated) and indirect (unconjugated) bilirubin will be ordered if total bilirubin > 5X ULN, Blood urea nitrogen (BUN or urea), Calcium, Chloride, Cholesterol, Creatinine, serum, Glucose, fasting plasma, Lactate dehydrogenase (LDH), Magnesium, Phosphorus, Potassium, Protein, total, Sodium, Triglycerides, Uric acid Urinalysis, Blood, Glucose, Ketones, Leukocyte esterase, pH, Protein Laboratory tests were graded using the National Cancer Institute-Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0 criteria
Time Frame: Assessed from day 1 up to within 30 days of last dose (Approximately 42 months)
Population: All treated participants
Measure: Number; unit: Number of abnormalities
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 52 | 7
Number of abnormalities
  Albumin | 0 | 0
  Alkaline Phosphatase (ALP) | 2 | 0
  Alanine Aminotransferase (ALT) | 1 | 0
  Aspartate Aminotransferase (AST) | 1 | 0
  Cholesterol, Total (TC): number analyzed (Participants) | 50 | 7
  Cholesterol, Total (TC) | 0 | 0
  Creatinine | 0 | 0
  Absolute Neutrophil Count | 0 | 0
  Hemoglobin | 0 | 0
  Lymphocytes (absolute) | 4 | 0
  Magnesium , serum: number analyzed (Participants) | 51 | 7
  Magnesium , serum | 0 | 0
  Neutrophils (absolute): number analyzed (Participants) | 51 | 7
  Neutrophils (absolute) | 0 | 0
  Glucose, fasting plasma: number analyzed (Participants) | 43 | 7
  Glucose, fasting plasma | 6 | 1
  Phosphorus, inorganic: number analyzed (Participants) | 51 | 7
  Phosphorus, inorganic | 0 | 0
  Platelet count | 2 | 0
  Bilirubin, total | 0 | 0
  Triglycerides: number analyzed (Participants) | 37 | 7
  Triglycerides | 0 | 0
  Triglycerides, fasting: number analyzed (Participants) | 42 | 7
  Triglycerides, fasting | 0 | 0
  Uric acid: number analyzed (Participants) | 51 | 7
  Uric acid | 3 | 0
  Leukocytes | 0 | 0

7. Secondary Outcome: Treatment Failure Rate (TFR)
Description: The TFR was to be calculated as the total number of subjects who discontinued the treatment for any reason (including disease progression, treatment toxicity, and death) at 24 weeks divided by the total number of subjects randomized/assigned to the arm and treated. In the monotherapy arm, the TFR was to be assessed while subjects were on monotherapy.
Time Frame: 24 weeks after initiation of study treatment
Population: TFR data was not collected for any participants because the study was terminated
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Changes in Absolute Copy Numbers and Relative Expression of Insulin Receptor Isoform A (IR-A) in Tumor Tissue in Response to Treatment
Description: Absolute copy numbers and relative expression of insulin receptor isoforms (IR-A, IR-B) in pre- and posttreatment fresh tumor tissues were to be measured. This outcome was not measured due to early termination of the study.
Time Frame: 24 weeks after initiation of study
Population: Data for this Outcome Measure was not collected for any participants because the study was terminated
Arm/Group | BMS 100 + LET | BMS 100
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to within 30 days of last dose (Approximately 42 months)
Description: AEs were collected starting at study medication administration on Day 1 and stopped at 7 days after the participant discontinued study medication or 7 days after the End of Treatment visit, if the visit occured at a later time
Arm/Group | BMS 100+LET | BMS 100
All-Cause Mortality (participants affected / at risk) | 5/52 | 0/7
Serious Adverse Events (participants affected / at risk) | 11/52 | 1/7
Other Adverse Events (participants affected / at risk) | 51/52 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 100+LET (N=52) | BMS 100 (N=7)
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Contrast Media Reaction (Injury, poisoning and procedural complications) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 100+LET (N=52) | BMS 100 (N=7)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 25 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 21 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 18 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Polydipsia (Metabolism and nutrition disorders) | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 28 | 4
Diarrhoea (Gastrointestinal disorders) | 20 | 3
Constipation (Gastrointestinal disorders) | 13 | 0
Vomiting (Gastrointestinal disorders) | 11 | 1
Dry Mouth (Gastrointestinal disorders) | 7 | 1
Abdominal Pain (Gastrointestinal disorders) | 5 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 34 | 3
Pyrexia (General disorders) | 5 | 0
Pain (General disorders) | 3 | 1
Asthenia (General disorders) | 3 | 0
Oedema Peripheral (General disorders) | 3 | 0
Gait Disturbance (General disorders) | 1 | 1
Peripheral Swelling (General disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 16 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 12 | 3
Dizziness (Nervous system disorders) | 10 | 2
Dysgeusia (Nervous system disorders) | 5 | 1
Neurological Symptom (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 3 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Weight Decreased (Investigations) | 15 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 0
Blood Creatinine Increased (Investigations) | 4 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 0
Platelet Count Decreased (Investigations) | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 0
Mucosal Infection (Infections and infestations) | 1 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 7 | 1
Anxiety (Psychiatric disorders) | 6 | 0
Vision Blurred (Eye disorders) | 7 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Polyuria (Renal and urinary disorders) | 4 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0
Menopausal Symptoms (Reproductive system and breast disorders) | 6 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 3 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1
Hot Flush (Vascular disorders) | 5 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.